CLINICAL TRIAL: NCT04784013
Title: Very High Power Ablation in Patients With Atrial Fibrillation Scheduled for a First Pulmonary Vein Isolation: the POWER-PLUS Study
Brief Title: Very High Power Ablation in Patients With Atrial Fibrillation Scheduled for a First Pulmonary Vein Isolation
Acronym: POWER-PLUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Prof. Dr. Mattias Duytschaever, Principal Investigator, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2800
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional group (Active Comparator)
  Interventions: Procedure: Conventional CLOSE-guided pulmonary vein isolation
- 90W-group (Active Comparator)
  Interventions: Procedure: High power short duration pulmonary vein isolation

INTERVENTIONS:
Procedure: Conventional CLOSE-guided pulmonary vein isolation — Point-by-point RF delivery will be performed aiming for a contiguous circle enclosing the veins. RF will be delivered in a temperature and flow-controlled mode (QMODE, target temperature 45°C, low flow temperature 40°C, cut-off temperature 50°C) with a power of 35W(posterior)/50W(anterior) (irrigation flow at 4-15ml/min). RF will be delivered until an ablation index (AI) of ≥400 at the posterior wall/roof/south pole and ≥550 at the anterior wall.
  Arms: Conventional group
Procedure: High power short duration pulmonary vein isolation — Point-by-point RF delivery will be performed aiming for a contiguous circle enclosing the veins. RF will be delivered in temperature-controlled mode (QMode+, target temperature 55°C, cut-off temperature 65°C) with a power of 90W (irrigation flow at 2-8ml/min). RF will be delivered for 4 sec at both the posterior and anterior wall.
  Arms: 90W-group

SUMMARY:
This prospective, randomized, controlled, unblinded, multicenter study aims at comparing procedural time between conventional CLOSE-guided pulmonary vein isolation (PVI) (35W/50W) versus very high power radiofrequency delivery (90W) in atrial fibrillation patients scheduled for a first PVI.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients scheduled for a first PVI only for paroxysmal atrial fibrillation (AF) (self-terminating or <7days) or persistent AF (persistent AF is defined as having an AF episode >7d); (patients with paroxysmal AF or short-standing persistent AF presenting with flutter, who are in need of a cavotricuspid isthmus ablation, are allowed to participate in this trial)
* Patients willing to sign informed consent

Exclusion Criteria:

* Patients with long-standing persistent AF (long-standing persistent AF is defined as having an AF episode >1yr)
* Previous ablation for AF
* Left atrium antero-posterior diameter >50 mm (parasternal long axis view, PLAX)
* AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
* Left atrial appendage (LAA) thrombus. LAA thrombus can be determined by preprocedural imaging: CT, transesophageal echocardiography or MRI.
* Left ventricular ejection fraction <35%.
* Cardiac surgery within the previous 90 days.
* Expecting cardiac transplantation or other cardiac surgery within 180 days.
* Coronary percutaneous transluminal coronary angioplasty/stenting within the previous 90 days or myocardial infarction within the previous 60 days.
* Documented history of a thromboembolic event within the previous 90 days.
* Diagnosed atrial myxoma.
* Significant restrictive, constrictive, or chronic obstructive pulmonary disease with chronic symptoms.
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment
* Women who are pregnant or who plan to become pregnant during the study.
* Acute illness or active infection at time of index procedure
* Advanced renal insufficiency
* Unstable angina.
* History of blood clotting or bleeding abnormalities.
* Contraindication to anticoagulation.
* Life expectancy less than 1 year.
* Presence of a condition that precludes vascular access.
* Unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Procedural time | Procedure (At time of ablation)
  Comparison of the procedural time (in minutes) between groups

SECONDARY OUTCOMES:
Single procedure atrial tachyarrhythmia freedom between months 4, 5 and 6 after the index ablation | Months 4-6 after ablation
  Atrial tachyarrhythmia will be monitored by Holter
Radiofrequency (RF) ablation time | Procedure (At time of ablation)
  Comparison of the RF ablation time (in seconds) between groups
Fluoroscopy dose | Procedure (At time of ablation)
  Comparison of the fluoroscopy dose (Gy cm²) between groups
First pass isolation rate | Procedure (At time of ablation)
  Reconnection of the veins after adenosine injection or waiting time

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Duytschaever, MD, PhD, Principal Investigator — AZ Sint-Jan AV
Locations (4):
- Medical University Hospital Graz, Graz, Austria
- AZ Sint-Jan Brugge-Oostende AV, Bruges, Please Select, Belgium
- UMC Leiden, Leiden, Netherlands
- Luzerner Kantonsspital, Lucerne, Switzerland

REFERENCES:
- [Derived] O'Neill L, El Haddad M, Berte B, Kobza R, Hilfiker G, Scherr D, Manninger M, Wijnmaalen AP, Trines SA, Wielandts JY, Gillis K, Lycke M, De Becker B, Tavernier R, Le Polain De Waroux JB, Knecht S, Duytschaever M. Very High-Power Ablation for Contiguous Pulmonary Vein Isolation: Results From the Randomized POWER PLUS Trial. JACC Clin Electrophysiol. 2023 Apr;9(4):511-522. doi: 10.1016/j.jacep.2022.10.039. Epub 2023 Jan 18. PMID 36752467